CLINICAL TRIAL: NCT03815201
Title: Effects of a Combined Physical Training and Protein Supplementation Intervention on Muscle Mass, Functional and Cognitive Performance, and Health-related Quality of Life in the Elderly: a Randomized Controlled Trial.
Brief Title: Protein Supplementation and Muscle Function in the Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Basque Health Service (Other Government)
Collaborators: University of the Basque Country (UPV/EHU) (Other); Hospital Universitario de Álava (Other)
Responsible Party: Principal Investigator, Ariadna Besga, Principal Investigator, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BasqueHS
Record Dates: First submitted 2019-01-15; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Sarcopenia
Keywords: muscle mass; protein supplementation; leucine; elderly; exercise training
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Placebo Comparator): exercise training program: 2 non-consecutive days per week during 12 weeks plus placebo ingestion post-training
  Interventions: Other: Group 1
- Group 2 (Active Comparator): exercise training program: 2 non-consecutive days per week during 12 weeks plus leucine-enriched protein supplementation post-training
  Interventions: Dietary Supplement: Group 2

INTERVENTIONS:
Dietary Supplement: Group 2 — leucine-enriched protein supplementation during the first 1/2 hour post-training
  Arms: Group 2
Other: Group 1 — placebo, an energy-matched mixture, during the first 1/2 hour post-training
  Arms: Group 1

SUMMARY:
Sarcopenia is a geriatric syndrome associated with functional lost and disability, leading to an increase in healthcare costs. Physical activity, especially multicomponent exercise program, seems to be the most effective intervention to delay disability in elderly patients.

The main objective of the current study is to determine if leucine-enriched protein ingestion after exercise training helps to increase muscle mass gains. Secondary outcomes will be to analyse the different effects among cognitive performance, depressive symptoms, disability, inflammation, quality of life and use of healthcare services.

A randomized controlled trial will be carried out to assess the objectives of the current study. Participants will be randomized into two different groups (N=40, each one): an exercise training control group and exercise training plus leucine-enriched protein ingestion intervention group. Exercise training will take 12 weeks of supervised training intervention and 12 weeks of non-supervised training intervention for both groups. Biological samples will be analysed in Biodonostia Health Research Institute and in the University of the Basque Country (UPV/EHU).

DETAILED DESCRIPTION:
Study protocol: Acute hospitalised, community-dwelling elderly patients will be recruited at internal medicine service of the Araba University Hospital (HUA). Patients that fulfil eligibility criteria for the study will be evaluated during their hospitalization for different aspects (Hospital Evaluation): handgrip, nutritional assessment using Mini Nutritional Assessment- Short Form Test (MNA-SF), functional assessment by Short Physical Performance Battery (SPPB), cognitive assessment (Pfeiffer test) and frailty assessment (Fried test). Once hospital evaluation is assessed patients will be offered to participate in the study. In case patients accept to participate, another assessment will be carried out on discharge date (Discharge Day Evaluation): handgrip, functional assessment (SPPB), 30-Second Chair Stand Test, 30-Second Arm Curl Test, the Timed Up ang Go (TUG) Test, 8 Foot Up and Go (FUG) Test, Gait Speed Test for 4- meters and for 8-meters. Patients will also take two accelerometers, a wrist accelerometer and a hip accelerometer, for a week.

A week after discharge day, patients will again be evaluated (Laboratory 1 (Lab 1) evaluation day): the same tests of discharge day will be repeated plus Berg Scale and 6-Minute Walking Test. Then, patients will wait until a group of 5-6 participants is formed. As soon as patients accept to participate, and when all evaluation tests involved until Lab 1 evaluation day are completed, participants will be randomized into two different groups: exercise training plus placebo control group (Group 1) and exercise training plus leucine-enriched protein ingestion intervention group (Group 2).

Participants will be called by telephone a week before the intervention starts for psychological assessment, blood analysis and Dual Energy X-ray Absorptiometry (DEXA) assessment.

The first day of intervention program all participants will be evaluated for nutritional assessment: Mini Nutritional Assessment (MNA) Test, a quantitative score (14-item) of adherence to the Mediterranean diet (Prevention with Mediterranean Diet (PREDIMED) questionnaire), two non-consecutive 24-hour dietary recall and anthropometry.

Exercise training intervention will be divided into supervised intervention and non-supervised intervention for both groups. Supervised intervention program will take 12 weeks and participants will have to assist 2 non-consecutive days per week to hospital for 1-hour exercise training. After those 12 weeks participants will take two accelerometers, a wrist accelerometer and a hip accelerometer, for a week. After that week participants will have to assist 2 non-consecutive days on the same week to complete: the same physical tests of Lab 1 evaluation day, anthropometry and nutritional tests, blood analysis and DEXA assessment. Individualised physical exercise recommendations will be explained and given to participants for the following 12 weeks of non-supervised intervention. During those weeks of non-supervised intervention, telephone monitoring will be made every two weeks.

When completing the study, at week 24, participants will be called by telephone to come to hospital for blood analysis, psychological assessment, nutritional tests and one 24-hour dietary recall, and to take the two accelerometers for a week. After a week, participants will be evaluated for physical assessment (the same physical tests of Lab 1 evaluation day will be carried out) and a second 24-hour dietary recall and anthropometry will be assessed.

The placebo and leucine-enriched protein supplementation will only be taken during supervised training period twice a week after 1-hour exercise training is completed. Participants will ignore what the supplement is, as the mixtures will be codified.

Protein supplementation will consist on 20gr of whey protein (a commercial preparation of Davisco®: BiPRO all-natural whey protein isolate) enriched with 3g of leucine (commercially prepared by Nutricia), and protein mixture will be diluted with 100ml of water. The placebo will be an energy-matched mixture.

The samples will be store at the Basque Biobank and then will be send to Biodonostia Health Research Institute for their analysis.

Sample size: power calculation has been done for the main variable: muscle mass increase. If 35 people are recruited on each group, a difference of unless 1.5 to 2kg will be detected in muscle mass with a standard deviation of 1.5-1.7kg and >80% of power, and an alfa level of 0.05. Taking into account that mortality can be about 30%, 40 participants will be recruited for each group.

Statistical analysis: variance analysis will be used to analyse the continuous variables and the Chi-square test for the categorical variables, both analyses will be used for the cross-cutting analysis. To evaluate the training effect on the primary and secondary variables general linear models will be used. Age and the pre-intervention value of any primary or secondary variable will be considered as covariates. The effect size and the statistical significance level for each of these effects will be calculated: group effect (between subjects), time effect (intra-subjects) and group*time interaction. Other possible interactions between group*sex and all other variables of the study will be determined. The analyses will be adjusted by multiple comparison test and the intend to treat principle will be applied for all analyses. For the analysis of missing data, such as for the participants that drop out from the program or did not meet the study criteria, different imputation methods will be used, and sensitivity analysis will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 70 years
* Punctuation at the Mini Mental State Questionnaire (MMSE): > or = 20.
* Any patient that fulfill the European Working Group on Sarcopenia in Older People (EWGSOP) criteria for sarcopenia diagnosis.
* Anyone who is able to walk alone, to walk using a walking stick or a walking frame, or to walk using parallel walking bars.
* Anyone able to understand the instructions or what is being said.
* Anyone signing the informed consent.

Exclusion Criteria:

* Chronic kidney disease
* To have suffered a heart attack in the last 3 months.
* To be unable to walk.
* To have suffered any fracture of the upper or lower limbs in the last 3 months.
* Anyone suffering from severe dementia.
* Autoimmune neuromuscular disorders (for example, myasthenia gravis, Guillain-Barré syndrome, inflammatory myopathies) or amyotrophic lateral sclerosis.
* Anyone refusing to sign the informed consent, or anyone who does not agree to the study protocol.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
muscle mass change | change from baseline muscle mass assessment to 12 weeks of supervised intervention
  muscle mass measured using dual-energy x-ray absorptiometry method

SECONDARY OUTCOMES:
Physical fitness change | change from baseline assessment to 12 weeks of supervised intervention and to the end of the study (at 6 months)
  combination of different tests to assess physical fitness

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna Besga, Principal Investigator — Basque Health Service
Locations (1):
- Hospital Santiago Apostol, Vitoria-Gasteiz, Alava, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR